CLINICAL TRIAL: NCT06422910
Title: Development and Investigation of the Effectiveness of Video Exercise Mobile Application for People With Knee Osteoarthritis
Brief Title: Video Exercise Mobile Application for People With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Ozden (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Tubitak diz OA
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Telerehabilitation; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Other: Telerehabilitation
- Control Group (Active Comparator)
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — Home exercises will be delivered through a video mobile application. In this application, exercises for knee osteoarthritis will be presented according to their types (stretching, strengthening, etc.). Videos deemed appropriate by the physiotherapist will be added to the exercise prescription and sent to the patients via message. Patients will have the opportunity to remotely access their own exercise prescription with visual, auditory and written commands.
  Translated with DeepL.com (free version)

SUMMARY:
The aim of our study is to realize an exercise training and follow-up system that individuals with knee OA can easily adapt.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary knee osteoarthritis (OA) according to the American College of Rheumatology (ACR) criteria
* Be qualified to use the mobile application and agree to use the application

Exclusion Criteria:

* Individuals with poor cognitive function or inadequate reading skills
* Individuals with neurological disorders that may affect mobility skills
* Individuals who have undergone knee joint surgery and individuals with traumatic injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Change from Baseline VAS at 8 weeks
  On a 0 cm straight line or numeric scale, the patient is asked to mark the pain they feel (0: no pain, 10: excruciating pain).
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline WOMAC at 8 weeks
  WOMAC consists of 3 main headings: pain intensity, stiffness and physical function. The total score ranges from 0 (no disability) to 96 (complete disability).
Satisfaction and expectation assessment | Change from Baseline Satisfaction and expectation assessment at 8 weeks
  On a 0 cm straight line or numeric scale, the patient will be asked to mark their pre-treatment expectation and post-treatment satisfaction level. 0 will represent the lowest expectation and satisfaction and 10 the highest expectation or satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Study Chair — Muğla Sıtkı Koçman University; Baki Umut Tuğay, PhD, Study Director — Muğla Sıtkı Koçman University; Barış Ethem Süzek, PhD, Principal Investigator — Muğla Sıtkı Koçman University; Nazan Tuğay, PhD, Principal Investigator — Sanko University; Zübeyir Sarı, PhD, Principal Investigator — Marmara University; İrem Çetinkaya, MSc, Principal Investigator — Haliç University; Gülser Cinbaz, MSc, Principal Investigator — İstanbul Medeniyet University
Locations (1):
- Fethiye State Hospital, Muğla, Fethiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozden F, Tugay BU, Coban O, Suzek BE, Tugay N, Sari Z, Cetinkaya I, Cinbaz G, Tumturk I. Development of video exercise-based mobile application to improve the clinical outcomes in patients with knee osteoarthritis: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Dec 27;18(1):39. doi: 10.1186/s13102-025-01503-w. PMID 41456047